CLINICAL TRIAL: NCT00422110
Title: A Phase IIb/III, Double-blind, Parallel-group, Placebo-controlled, Randomized Study: Evaluation of the Efficacy and Safety of Seletracetam as Adjunctive Treatment in Subjects (≥16 to 70 Years Old) With Refractory Partial Onset Seizures.
Brief Title: A Study to Evaluate the Efficacy and Safety of Seletracetam in Adult Patients With Refractory Partial Onset Seizures
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N01272
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Epilepsies, Partial
Keywords: Seletracetam; Epilepsies; Partial; Epilepsy; Focal
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy | interventions — Seletracetam

INTERVENTIONS:
Drug: Seletracetam

SUMMARY:
This study will evaluate the effectiveness and safety of seletracetam when it is used in addition to other anti-epileptic medications by patients with partial onset seizures. It will also help to determine the best dose to use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from 16 to 70 years old
* Confirmed diagnosis of focal epilepsy
* Partial seizures uncontrolled while taking 1 or 2 AEDs
* At least 8 partial seizures during the 8-week baseline period

Exclusion Criteria:

* Seizures occurring only in clusters
* Status epilepticus within 1 year
* Progressive CNS disorder
* Other serious or uncontrolled diseases

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-05

PRIMARY OUTCOMES:
Evaluate the efficacy of seletracetam compared to placebo in reducing seizure frequency in subjects with partial onset seizures not fully controlled despite treatment with 1 - 2 concomittant AEDs

SECONDARY OUTCOMES:
Explore the dose/clinical response relation; safety and tolerability; effects of treatment on patients' Health-Related Quality of Life (HRQoL)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Bennett, PhD, Study Director — UCB Pharma